CLINICAL TRIAL: NCT00937248
Title: A Randomized Study Evaluating Set-up Reproducibility Using Cone Beam CT (CBCT) With and Without a Customized Vacuum Immobilization Device (CVID) in Rectal Cancer Patients Treated With Preoperative Pelvic Radiation Therapy
Brief Title: Cone Beam Computed Tomography (CT) (CBCT) With and Without a Customized Vacuum Immobilization Device (CVID)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: UHN REB 09-0086-CE
Record Dates: First submitted 2009-07-08; First posted 2009-07-10 (Estimated); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Rectal Cancer
Keywords: Cone Beam CT in rectal cancer patients; Immobilizing rectal cancer patients; Image guided radiotherapy in rectal cancer patients
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Interventional (Experimental): Patient randomized to be immobilized using a prone pillow and simple ankle fixation device with a CVID.
  Interventions: Device: Customized Vacuum Immobilization Device (CVID)
- Standard Arm (Active Comparator): Patient randomized to be immobilized using a prone pillow and simple ankle fixation device without a CVID
  Interventions: Device: prone pillow and simple ankle fixation device

INTERVENTIONS:
Device: prone pillow and simple ankle fixation device — Patients will lie face down (prone) on a soft cushion made of foam under their face and upper chest. Additionally, there is a foam support placed at the ankles.
  Arms: Standard Arm
Device: Customized Vacuum Immobilization Device (CVID) — This device is a bean bag like cushion that is placed from the abdomen to the thighs. When a patient is comfortably lying on this device, air within the bag is suctioned out resulting in an impression or cast of a patient.
  Arms: Interventional

SUMMARY:
This study is designed to investigate whether or not the use of a customized vacuum immobilization device (CVID) to immobilize rectal cancer patients undergoing preoperative pelvic radiation therapy improves the positional stability of patients during each radiation treatment. This question is more relevant now in the era of image-guided radiation therapy (IGRT). Using state of the art IGRT technologies such as cone beam CT (CBCT) scanning, assessments of the accuracy of treatment delivery can be made during a course of radiation therapy allowing for patient set-up corrective strategies to be implemented. The use of CBCT scanning may minimize any potential benefit of of a CVID if the patient's pretreatment position can be corrected prior to treatment and our current immobilization strategy results in a stable patient position. While it is seemingly intuitive to assume that the use of CVID results in better patient stability, there is actually little data to support this.

DETAILED DESCRIPTION:
Rectal cancer accounts for 5% of all cancers diagnosed in Canada for both men and women between 1995 and 2004 (Public Health agency of Canada _ Health 2004). Preoperative radiotherapy (RT), with or without chemotherapy, is an accepted treatment for patients with locally advanced rectal carcinoma followed by surgical resection (Bosset and Horiot 2001; Sauer, Fietkau et al. 2003; Birgisson, Talback et al. 2005). The current standard treatment at Princess Margaret Hospital (PMH) is preoperative pelvic radiation therapy to a total dose of 50 Gy/25 fractions/5 weeks. The total radiation dose is reduced to 45 Gy/25 fractions/5 weeks when there is a concern about the volume of small bowel within the treatment volume. Radiation therapy is delivered with 5-fluorouracil (5-FU), 225mg/m2/24h, by protracted venous infusion (PVI) or oral capecitabine, 825 mg/m2 BID for 5 weeks, starting the first day and completing the day of last day of radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Any rectal cancer patient who is to receive a 5 week course of preoperative pelvic radiation therapy with or without concurrent chemotherapy
* Prone treatment position
* Age 18 years or older
* Informed consent

Exclusion Criteria:

* Inability to provide informed consent
* Inability to tolerate treatment in the prone position
* Pregnancy
* Patients with unilateral or bilateral metallic total hip replacements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-04; Primary Completion 2023-04-21 (Actual); Study Completion 2023-04-21 (Actual)

PRIMARY OUTCOMES:
Comparing the use of a prone pillow and simple ankle fixation device vs. the use of a CVID for immobilization rectal patients during the course of preoperative radiation therapy using KV CBCT for IGRT. | 2 years

SECONDARY OUTCOMES:
quantify interfractional set-up displacements using either of the two devices;determine a standard planning target volume margin; evaluate the role of soft-tissue image matching for IGRT using CBCT. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: John Kim, MD, Principal Investigator — University Health Network, Princess Margaret Hospital
Locations (1):
- University Health Network, Princess Margaret Hospital, Toronto, Ontario, Canada